CLINICAL TRIAL: NCT00604825
Title: A Parallel-group, Double-blind, Randomized, Placebo-controlled, Active Comparator, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Two Doses of GSK232802 Administered Orally as Monotherapy for 12 Weeks in Healthy Postmenopausal Women With Moderate to Extremely Severe Vasomotor Symptoms
Brief Title: Treatment Of Hot Flashes/Flushes In Postmenopausal Women (WARM Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105106
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Menopausal and Female Climacteric States
Keywords: menopause; hormone therapy; hot flashes; vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Other: Placebo
- GSK232802 (Active Comparator): GSK232802
  Interventions: Drug: GSK232802
- PREMARIN (Experimental): PREMARIN
  Interventions: Drug: PREMARIN

INTERVENTIONS:
Drug: Other: Placebo
  Arms: Placebo
Drug: GSK232802
  Arms: GSK232802
Drug: PREMARIN
  Other Names: Other: Placebo; GSK232802
  Arms: PREMARIN

SUMMARY:
The purpose of this study is to determine whether GSK232802 is safe and effective in reducing the frequency and severity of hot flashes associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Postmenopausal women aged 40 to 65 years old; postmenopausal defined as:

  i.Amenorrheic for at least 12 consecutive months* OR ii.At least 6 weeks post-surgical bilateral oophorectomy† with or without hysterectomy.

  *Note: Although duration of amenorrhea is initially determined by subject history at the time of the screening visit (Visit 1), menopausal status must be confirmed by demonstrating levels of follicle stimulating hormone (FSH) >40 mIU/mL (SI: >40 IU/L) and estradiol <35pg/mL (SI: <128pmol/L) at entry. Screening reports provided by the Central Laboratory must be carefully reviewed to determine menopause eligibility prior to conducting Visit 2 assessments. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or estradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility should be discussed with the study medical monitor.

  †For women who are surgically menopausal, a copy of the pathology report or a statement on letterhead from the subject's physician documenting both ovaries have been removed or biochemical evidence of post-menopausal status as noted above is required prior to conducting Visit 2 assessments.
* A minimum average frequency of seven daily moderate to extremely severe hot flashes or episodes of night sweats sufficient to cause the patient to seek treatment (these episodes must be documented during the baseline period and the subject must have recorded frequency and severity of symptoms for a minimum of eight days in order to be eligible for randomization). This average frequency will be calculated by summing the number of moderate, severe, and extremely severe VMS events during the baseline period and dividing by the total number of non-missing days during this period, with details related to the definition of non-missing days described in Section 6.3.1.
* BMI within the range 19 to 35 kg/m2, inclusive.
* Subject has provided signed and dated written informed consent before admission to the study.
* Subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Investigator considers subject unfit for the study as a result of medical history, physical examination, or screening tests.
* Use of prescription or non-prescription drugs including:

  i.Hormone therapy (estrogen or estrogen/progestin combination or related products) within the following time period prior to conduct of Visit 1 assessments:
* 4 weeks for prior vaginal hormonal products (rings, creams, gels) or transdermal estrogen or estrogen/progestin products.
* 4 weeks for oral estradiol (e.g., micronized estradiol) or SERM products (e.g., raloxifene).
* 8 weeks for prior oral conjugated (equine or synthetic) estrogen or estrogen/progestin products or for prior intrauterine progestin therapy.
* 3 months for prior progestin implants or injectable estrogen.
* 6 months for prior estrogen pellet therapy or injectable progestin. ii.Use of putative therapies for VMS relief (e.g., selective serotonin reuptake inhibitors [SSRIs], serotonin-norepinephrine reuptake inhibitors [SNRIs], clonidine, gabapentin, tibolone, methyldopa, and the phytoestrogens black cohosh and red clover) within the past 30 days or 5 half-lives (whichever is longer) prior to conduct of Visit 1 assessments (note: half-lives will be provided in the SPM). Use of non-medication treatments for VMS, such as acupuncture and biofeedback, and other complementary or alternative therapies for VMS relief (with the exception of black cohosh and red clover which require a specified washout previously noted) must be discontinued at Visit 1.

iii.Use of weight loss drugs (e.g., phentermine, sibutramine, orlistat, rimonabant) within 3 months of the first dose of investigational product. Other complementary or alternative therapies for weight reduction must be discontinued at Visit 1. See SPM for listing.

iv.Use of pravastatin [Pravachol/Lipostat], rosuvastatin [Crestor], or pitavastatin [Livalo] within the past 30 days or 5 half-lives (whichever is longer) of the first dose of investigational product (note: half-lives will be provided in the SPM. Uses of other statins, for example simvastatin [Zocor], atorvastatin [Lipitor], fluvastatin [Lescol], lovastatin [Mevacor] is allowed).

v.Use of bupropion, orphenadrine [Norflex], cyclophosphamide, efavirenz, ifosfamide, or methadone (because of the potential for GSK232802 to inhibit CYP2B6), or use of paclitaxel, torsemide, amodiaquine, repaglinide, rosiglitazone, or pioglitazone (because of the potential for GSK232802 to inhibit CYP2C8) within the past 30 days or 5 half-lives (whichever is longer) of the first dose of investigational product (note: half-lives will be provided in the SPM).

Please note: Regardless of the reason for prescribing, use of the medications and therapies defined within Exclusion 2 above is prohibited. Concurrent administration of anti-depressants, anti-hypertensives, lipid-lowering therapies, etc. not specifically excluded above is allowed. See SPM for detailed listings and relevant half lives.

- Use of investigational drug within the past 30 days or 5 half-lives (whichever is longer) before the first dose of investigational product.

* Uterine disease or medical condition including:
* Bi-layer endometrial thickness greater than 5mm as determined by TVUS, or for women with a non-informative TVUS, a single layer thickness of greater than 3 mm determined by SIS; presence of fibroids that obscure evaluation of endometrium by TVUS;
* History of uterine cancer; evidence of endometrial hyperplasia or cancer as assessed by a screening endometrial biopsy. (Note: if a subject has insufficient tissue for diagnosis at screening, but bi-layer endometrial thickness by TVUS is ≤5mm or single wall thickness by SIS is ≤3mm, she may still be eligible for study entry if she meets the remaining inclusion/exclusion criteria);
* Evidence of an endometrial polyp with hyperplastic or malignant epithelium;
* Unexplained or unusual endometrial bleeding; or uterine surgery (other than hysterectomy*) within the past 6 months; *Note: hysterectomy must have been conducted at least 6 weeks prior to screening Visit 1. See also Inclusion criterion 1.
* Abnormal cervical Pap smear with evidence of cervical dysplasia greater than or equal to low grade squamous intraepithelial lesion (LSIL) or with a diagnosis of atypical squamous cells of undetermined significance (ASCUS) that is HPV High Risk positive, or glandular lesions including but not limited to atypical glandular cells of undetermined significance (AGUS), adenocarcinoma in situ (AIS) or malignancy
* History of breast or ovarian cancer. Any clinically significant findings on mammography suspicious of breast malignancy that would require additional clinical testing to rule out breast cancer (note: simple cysts confirmed by ultrasound are allowed).

Note: A screening mammogram is required unless the subject has had a mammogram performed within the last 12 months. If local mammography or medical management guidelines restrict the frequency with which mammograms can be performed, or impose age restrictions on the use of mammography, such that a subject may be unable to undergo the study-required screening mammogram, then these subjects must not be enrolled in the study. See Section 6.2.7.

- Cardiovascular conditions including: i. Systolic blood pressure (BP) outside the range 80 to 150 mmHg, diastolic BP outside the range 50 to 90 mmHg, and/or heart rate outside the range 40 to 100 bpm. Subjects with mild to moderate hypertension who are controlled on a stable antihypertension regimen may be enrolled if they meet the inclusion/exclusion criteria.

ii. Symptomatic or asymptomatic arrhythmia of any clinical significance. iii. Any clinically significant abnormality identified on the screening 12-lead ECG. Subjects with QTc prolongation (QTc interval >450msec) will be excluded.

iv. Has a documented history (within the last year) of myocardial infarction, angina, or has undergone coronary artery bypass surgery and/or percutaneous transluminal coronary angioplasty (PTCA).

v. History of venous or arterial thromboembolic disease (e.g., deep vein thrombosis, pulmonary embolism, stroke), history of known coagulopathy or abnormal coagulation factors; increased thrombotic risk as evidenced by positive APC resistance (APCR) evaluated at screening.

- Has a documented history of hepatobiliary disease or hepatic enzyme elevation including any one of the following: i.ALT or direct (conjugated) bilirubin values 1.5-fold higher than the ULN at screening.

ii.Fasting triglycerides >400mg/dL (SI: >4.52mmol/L) at screening. If a subject is receiving a lipid-lowering therapy, then she must be on a stable dose for at least 1 month before screening.

* Has an abnormal thyroid function test assessed by TSH at screening (TSH <0.1uU/mL or >10uU/mL [SI: <0.1mU/L or >10mU/L] ).

Note: If the TSH is mildly out of range at screening (TSH < 15U/mL), the subject may have her dose adjusted (if already on exogenous therapy) or have therapy initiated as deemed appropriate by the subject's physician, followed by a 3-4 week period to allow adequate equilibration. The TSH may then be re-assayed for eligibility purposes after this stabilization period has been completed. The subject should not progress through subsequent V2 assessments until re-assay demonstrates the TSH is within acceptable protocol-defined limits. Subjects with suppressed levels of TSH, <0.1U/mL, may have dose adjustment if free T4 is in normal range, and they are on exogenous thyroxine therapy.

* Has either a previous disease or current medical condition, which as judged by the investigator, may affect the interpretation of efficacy or safety data or which otherwise contraindicates participation in a clinical study with a new chemical entity. These diseases include, but are not limited to, cardiovascular disease, malignancy*, complex ovarian pathology, hepatic disease, renal disease, hematological disease, neurological disease, or endocrine disease. A subject with diabetes may be included if her diabetes is well controlled (i.e., HbA1c level is less than 8% at screening).

  *Note: Any history of malignancy within the past 5 years is exclusionary with the exception of basal cell (excluded if within the prior 2 years) or squamous cell (excluded if within the prior one year) carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible. Note that this timeframe does not apply to uterine, breast, and ovarian cancers which are defined in Exclusions 4 and 5 above.
* History of alcohol or substance abuse or dependence in the 12 months before screening as determined by the investigator.
* Positive results for hepatitis B surface antigen or hepatitis C antibodies as evaluated at screening Visit 1. Known history of HIV.
* Donation of blood in excess of 500mL within a 56-day period before screening.
* History or presence of allergy to the investigational product or drugs of this class (e.g., raloxifene), or history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2007-07-17 (Actual); Primary Completion 2008-07-23 (Actual); Study Completion 2008-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (38):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Crystal River, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Hilton Head Island, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
- Argentina (4):
  - GSK Investigational Site, Buenos Aries, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (5):
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Dulwich, South Australia
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Subiaco, Western Australia
- Germany (11):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mühlheim am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Nordhausen, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (4):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Florence, Tuscany
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Wellington
- Spain (3):
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Santiago de Compostela
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Kungsbacka
  - GSK Investigational Site, Uddevalla
- United Kingdom (6):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Waterloo, Liverpool

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from at 75 centers (2 in Spain, 3 each in Argentina, New Zealand and the United Kingdom, 4 in Italy, 5 in Australia, 6 in Sweden, 12 in Germany, and 37 in the United States) from 17-July-2007 to 23-July-2008.
Pre-assignment Details: A total of 982 healthy postmenopausal participants with moderate to extremely severe vasomotor symptoms were screened (626 screen failures) and 356 were randomized.
Groups:
- Placebo: Eligible participants received placebo tablets/capsules to match GSK232802 tablets and Premarin capsules, one tablet or capsule via oral route at approximately the same time each morning for a total period of 12 weeks.
- GSK232802 25 mg: Eligible participants received GSK232802 25 milligram (mg) tablets, one tablet via oral route at approximately the same time each morning for a total period of 12 weeks.
- GSK232802 75 mg: Eligible participants received GSK232802 75 mg tablets, one tablet via oral route at approximately the same time each morning for a total period of 12 weeks.
- Premarin 0.3 mg: Eligible participants received Premarin 0.3 mg capsules, one capsule via oral route at approximately the same time each morning for a total period of 12 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Started | 90 | 87 | 89 | 90
Completed | 81 | 72 | 73 | 79
Not Completed | 9 | 15 | 16 | 11
Not completed — Adverse Event | 2 | 6 | 7 | 4
Not completed — Lost to Follow-up | 0 | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 5 | 5
Not completed — Lack of Efficacy | 3 | 2 | 1 | 0
Not completed — Did not meet eligibility criteria | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Exclusion criterion met | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK232802 25 mg: Eligible participants received GSK232802 25 mg tablets, one tablet via oral route at approximately the same time each morning for a total period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg | Total
Number analyzed (Participants) | 90 | 87 | 89 | 90 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (4.17) | 54.9 (4.72) | 54.2 (4.78) | 54.0 (5.18) | 54.6 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 87 | 89 | 90 | 356
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 9 | 9 | 9 | 31
  White | 84 | 78 | 79 | 79 | 320
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) and Number of Participants With Mild, Moderate and Severe AE
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. The severity of AEs was assessed by the investigator as mild, moderate or severe.
Time Frame: Up to 21 weeks
Population: Safety Population which comprised of all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Participants
  AE | 54 | 52 | 45 | 51
  SAE | 2 | 0 | 1 | 1
  Mild AE | 19 | 20 | 8 | 18
  Moderate AE | 30 | 25 | 32 | 23
  Severe AE | 5 | 7 | 4 | 10

2. Primary Outcome: Change From Baseline in Vital Signs of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 12
Description: SBP and DBP were measured after the participant had rested for at least 5 minutes in a sitting or supine position. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline in SBP and DBP at Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Millimeters of mercury
  SBP: number analyzed (Participants) | 81 | 72 | 74 | 79
  SBP | 2.6 (15.26) | 1.8 (12.19) | -1.6 (11.04) | -0.4 (12.61)
  DBP: number analyzed (Participants) | 81 | 72 | 74 | 79
  DBP | 0.1 (8.38) | 1.0 (9.28) | 0.7 (7.04) | -0.1 (9.06)

3. Primary Outcome: Change From Baseline in Vital Sign of Heart Rate at Week 12
Description: Heart rate was measured after the participant had rested for at least 5 minutes in a sitting or supine position. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline in heart rate at Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Beats per minute | -0.2 (9.84) | 0.6 (8.27) | 2.8 (8.09) | 0.3 (9.66)

4. Primary Outcome: Change From Baseline in Thyroid Stimulating Hormone (TSH) at Week 12
Description: Serum hormone markers included TSH. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline in TSH at Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliunits/Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 78
Milliunits/Liter | 0.236 (0.8942) | 0.034 (0.9951) | 0.397 (1.3453) | 0.238 (0.9280)

5. Primary Outcome: Change From Baseline in Thyroxine (T4) and Insulin at Week 12
Description: Serum hormone markers included T4 and additional pharmacodynamics marker included insulin. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline in T4 and insulin at Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomole per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Picomole per Liter
  T4: number analyzed (Participants) | 81 | 72 | 74 | 79
  T4 | -0.190 (1.8660) | -0.350 (1.6473) | -0.582 (1.6272) | -0.425 (1.8863)
  Insulin: number analyzed (Participants) | 79 | 71 | 73 | 74
  Insulin | 12.747 (83.3643) | 4.563 (49.2320) | 3.205 (44.1258) | -19.297 (137.5697)

6. Primary Outcome: Change From Baseline in Fasting Lipid Profile at Week 12
Description: Fasting lipids included total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholestereol direct and triglycerides. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline in fasting lipid profile at Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Millimole per Liter
  Cholesterol: number analyzed (Participants) | 81 | 71 | 73 | 79
  Cholesterol | 0.055 (0.7977) | 0.019 (0.5600) | -0.203 (0.5985) | -0.062 (0.7300)
  HDL cholestereol, direct: number analyzed (Participants) | 81 | 71 | 73 | 79
  HDL cholestereol, direct | 0.047 (0.1851) | 0.093 (0.2296) | 0.070 (0.2184) | 0.069 (0.2357)
  LDL cholesterol: number analyzed (Participants) | 81 | 70 | 71 | 79
  LDL cholesterol | 0.030 (0.6987) | -0.221 (0.4564) | -0.430 (0.5290) | 0.208 (0.6744)
  Triglycerides: number analyzed (Participants) | 81 | 71 | 73 | 79
  Triglycerides | -0.060 (0.7480) | 0.309 (0.4718) | 0.370 (0.6892) | 0.166 (0.4941)

7. Primary Outcome: Change From Baseline in Bi-layer Endometrial Thickness Measured by Transvaginal Ultrasound (TVUS) or Saline Infusion Sonohysterography (SIS)
Description: All participants with an intact uterus participating in this study underwent a TVUS at Baseline and at Week 12, to investigate the cause of any abnormal uterine bleeding during the study. In the event the TVUS was not well visualized or there were abnormal findings at either visit, or the bi-layer thickness exceeded 5 millimeter at Week 12, a SIS was conducted to visualize the anterior and posterior walls. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline and Week 12 in heart rate are presented.
Time Frame: Baseline (Week 0) to Week 12
Population: Uterine Safety Population which comprised of all randomized participants who had a uterus and also received at least one dose of investigational product. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 54 | 53 | 52 | 51
Millimeter
  TVUS Bi-layer Endometrial Thickness: number analyzed (Participants) | 48 | 44 | 43 | 45
  TVUS Bi-layer Endometrial Thickness | -0.07 (1.255) | 0.13 (1.383) | 0.79 (1.895) | 1.12 (2.051)
  SIS Posterior Endometrial Thickness: number analyzed (Participants) | 1 | 1 | 0 | 0
  SIS Posterior Endometrial Thickness | 8.40 (NA) — Single participant | 0.90 (NA) — Single participant |  |
  SIS Anterior Endometrial Thickness: number analyzed (Participants) | 1 | 1 | 0 | 0
  SIS Anterior Endometrial Thickness | -1.20 (NA) — Single participant | 1.70 (NA) — Single participant |  |
  SIS Total Endometrial Thickness: number analyzed (Participants) | 1 | 1 | 0 | 0
  SIS Total Endometrial Thickness | 7.20 (NA) — Single participant | 2.60 (NA) — Single participant |  |

8. Primary Outcome: Endometrial Biopsy Pathology
Description: Endometrial biopsies were conducted at Baseline and end-of-treatment (end-of-treatment values were defined as the last available post-Baseline values before treatment was stopped) for all study participants with an intact uterus. These procedures were performed by an experienced physician. Each biopsy was obtained after the TVUS was performed. Proliferative endometrium also meant hyperplasia without atypia (normal).
Time Frame: Baseline (Week 0) to Week 12
Population: Uterine safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 54 | 53 | 52 | 51
Participants
  Baseline: number analyzed (Participants) | 53 | 53 | 52 | 51
  Baseline: Normal | 29 | 33 | 34 | 31
  Baseline: No tissue/insufficient tissue | 23 | 19 | 17 | 20
  Baseline: Proliferative endometrium | 1 | 0 | 1 | 0
  Baseline: Progestational endometrium | 0 | 1 | 0 | 0
  Baseline: Polyp | 0 | 0 | 0 | 0
  End of treatment: number analyzed (Participants) | 42 | 47 | 40 | 45
  End of treatment: Normal | 19 | 27 | 24 | 31
  End of treatment: No tissue/insufficient tissue | 23 | 19 | 16 | 9
  End of treatment: Proliferative endometrium | 0 | 1 | 0 | 3
  End of treatment: Progestational endometrium | 0 | 0 | 0 | 1
  End of treatment: Polyp | 0 | 0 | 0 | 1

9. Primary Outcome: Occurrence of Withdrawal Bleeding-duration of Spotting/Bleeding
Description: After completion of the 12-week treatment period, participants with an intact uterus received a 14-day cycle of progestogen (10 mg medroxyprogesterone acetate [MPA]) to induce withdrawal bleeding. All participants were required to return to clinic for Follow-Up Visit. Participants were asked to record occurrence of bleeding/spotting each day, from the day MPA dosing began until Follow-up using the following criteria: None (no bleeding or spotting), Spotting: any vaginal flow requiring not more than one sanitary napkin or tampon per day (lightly stained and not soaked through) and Bleeding: any vaginal flow requiring more than one sanitary napkin or tampon per day. The following information was recorded in electronic case report form: start and stop date of MPA administration as well as dates of any spotting/bleeding. Duration of spotting or bleeding is presented.
Time Frame: Up to Follow-up (Day 112)
Population: Uterine Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 48 | 48 | 42 | 47
Days | 0.0 [0 to 23] | 0.0 [0 to 36] | 0.0 [0 to 45] | 1.0 [0 to 30]

10. Primary Outcome: Occurrence of Withdrawal Bleeding-number of Days of Spotting, Number of Days of Bleeding, Number of Days of Spotting/Bleeding Combined
Description: After completion of the 12-week treatment period, participants with an intact uterus received a 14-day cycle of progestogen (10 mg MPA) to induce withdrawal bleeding. All participants were required to return to clinic for Follow-Up Visit. Participants were asked to record occurrence of bleeding/spotting each day, from the day MPA dosing began until Follow-up using the following criteria: None (no bleeding or spotting), Spotting: any vaginal flow requiring not more than one sanitary napkin or tampon per day (lightly stained and not soaked through) and Bleeding: any vaginal flow requiring more than one sanitary napkin or tampon per day. The following information was recorded in electronic case report form: start and stop date of MPA administration as well as dates of any spotting/bleeding. Duration of spotting, bleeding and also spotting/bleeding combined is presented.
Time Frame: Up to Follow-up (Day 112)
Population: Uterine Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 48 | 48 | 42 | 47
Days
  Number of days of spotting | 0.0 [0 to 12] | 0.0 [0 to 9] | 0.0 [0 to 10] | 0.0 [0 to 16]
  Number of days of bleeding | 0.0 [0 to 5] | 0.0 [0 to 4] | 0.0 [0 to 5] | 0.0 [0 to 17]
  Number of days of spotting/bleeding combined | 0.0 [0 to 14] | 0.0 [0 to 11] | 0.0 [0 to 13] | 1.0 [0 to 20]

11. Primary Outcome: Mean Change in Frequency of Vasomotor Symptoms (VMS) From Baseline at Week 12
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an electronic diary (eDiary) using as Global Change Question. The frequency was assessed using the question 1 as "Since you started the study medication, how has the number of your hot flashes (including night sweats) changed?". the response was rated on a 7-point scale from +3 to -3, where +3=A great deal better, +2=Moderately better, +1=A little better, 0=No change, -1=A little worse, -2=Moderately worse and -3=A great deal worse. The score ranged from +3 to -3, where +3 implied absence of symptoms and lower score implied more severe symptoms. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Adjusted mean is presented as least square mean.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent-to-Treat Population (ITT) Population which comprised of all randomized participants. Last Observation Carried Forward (LOCF) was the imputation technique used.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale | -5.53 (0.466) | -4.78 (0.522) | -4.31 (0.500) | -7.59 (0.479)
Statistical Analysis 1: Comparison: Placebo vs GSK232802 25 mg; Placebo vs. GSK232802 25 mg; Test type: Superiority; p = 0.215, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = 0.75, 95% CI 2-sided [-0.44 to 1.93]
Statistical Analysis 2: Comparison: Placebo vs GSK232802 75 mg; Placebo vs. GSK232802 75 mg; Test type: Superiority; p = 0.041, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = 1.21, 95% CI 2-sided [0.05 to 2.37]
Statistical Analysis 3: Comparison: Placebo vs Premarin 0.3 mg; Placebo vs. Premarin 0.3 mg; Test type: Superiority; p < 0.001, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = -2.06, 95% CI 2-sided [-3.20 to -0.92]

12. Primary Outcome: Mean Change in Severity of VMS From Baseline at Week 12
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an eDiary using global change questions. VMS severity was as follows: mild=score of 1 (brief wave of heat with minimal discomfort, usually without perspiration; able to continue activity [or sleep]), moderate=score of 2(heat with some discomfort, usually with perspiration; minimal interruption of activity [or sleep]), severe=score of 3(intense heat with considerable discomfort, usually with heavy sweating; may be unable to resume activity [or sleep] right away) and extremely severe=score of 4 (unbearable heat with intense discomfort, usually with pouring sweat; may be unable to resume activity [or sleep] for quite a while). Total score ranged from 1 to 4 and is the sum of severity scores divided by total number of VMS events. Higher score indicates worst condition. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF analysis. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale | -0.37 (0.093) | -0.21 (0.104) | -0.05 (0.099) | -0.89 (0.095)
Statistical Analysis 1: Comparison: Placebo vs GSK232802 25 mg; Placebo vs. GSK232802 25 mg; Test type: Superiority; p = 0.202, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = 0.15, 95% CI 2-sided [-0.08 to 0.38]
Statistical Analysis 2: Comparison: Placebo vs GSK232802 75 mg; Placebo vs. GSK232802 75 mg; Test type: Superiority; p = 0.008, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = 0.31, 95% CI 2-sided [0.08 to 0.54]
Statistical Analysis 3: Comparison: Placebo vs Premarin 0.3 mg; Placebo vs. Premarin 0.3 mg; Test type: Superiority; p < 0.001, General linear model — Analysis included the terms for: Treatment + Baseline + country + uterine strata; Adjusted Mean Difference = -0.52, 95% CI 2-sided [-0.75 to -0.30]

13. Primary Outcome: Change From Baseline in Thrombotic Marker- Fibrinogen at Week 12
Description: Thrombotic marker included fibrinogen. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per LIter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 70 | 65 | 67 | 75
Gram per LIter | -0.081 (0.5889) | -0.246 (0.8377) | -0.293 (0.6487) | -0.198 (0.5291)

14. Primary Outcome: Change From Baseline in Thrombotic Marker- Tissue Plasminogen Activator (tPA) Antigen at Week 12
Description: Thrombotic marker included tPA antigen. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 79 | 70 | 70 | 75
Microgram per Liter | 0.200 (3.0996) | -0.139 (2.2818) | -1.224 (2.8039) | 0.115 (2.4548)

15. Primary Outcome: Change From Baseline and Week 12 in Inflammatory Marker- High Sensitivity C-reactive Protein (Hs-CRP) at Week 12
Description: Inflammatory marker included hs-CRP. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milligram per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 78 | 69 | 72 | 79
Milligram per Liter | 0.008 (1.5780) | 2.181 (9.4203) | 0.833 (2.3385) | 0.557 (3.6617)

16. Primary Outcome: Change From Baseline and Week 12 in Inflammatory Marker- Endothelin-1 at Week 12
Description: Inflammatory marker included Endothelin-1. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 76 | 67 | 71 | 73
Nanogram per Liter | -1.204 (1.4544) | -0.897 (1.3425) | -1.087 (1.5720) | -0.945 (1.6884)

17. Primary Outcome: Change From Baseline and Week 12 in Hematology Parameter- Hematocrit at Week 12
Description: Hematology parameter included hematocrit. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 76
Fraction | -0.003 (0.0303) | -0.006 (0.0192) | -0.019 (0.0313) | -0.002 (0.0198)

18. Primary Outcome: Change From Baseline in Hematology Parameter- Mean Corpuscle Hemoglobin (MCH) at Week 12
Description: Hematology parameter included MCH. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 76
Picograms | -0.260 (0.6118) | -0.221 (0.6094) | -0.207 (0.6878) | -0.326 (0.6005)

19. Primary Outcome: Change From Baseline in Hematology Parameter- Mean Corpuscle Volume (MCV) at Week 12
Description: Hematology parameter included MCV. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 76
Femtoliters | -0.813 (1.8356) | -0.169 (2.1179) | -0.694 (2.2558) | -0.368 (1.7802)

20. Primary Outcome: Change From Baseline in Hematology Parameter- Red Blood Cell (RBC) Count at Week 12
Description: Hematology parameter included RBC count. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 76
Trillion cells per Liter | 0.005 (0.3073) | -0.059 (0.1833) | -0.179 (0.3053) | -0.005 (0.2103)

21. Primary Outcome: Change From Baseline in Hematology Parameters- Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at Week 12
Description: Hematology parameters included Hemoglobin and MCHC. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 76
Gram per Liter
  Hemoglobin | -1.275 (8.9216) | -2.887 (5.6050) | -5.944 (8.3293) | -1.382 (6.3476)
  MCHC | -0.275 (8.2768) | -2.000 (9.0885) | 0.500 (11.1381) | -2.079 (8.0957)

22. Primary Outcome: Change From Baseline in Hematology Parameters- Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Segmented Neutrophils, Total Neutrophils and White Blood Cell (WBC) Count at Week 12
Description: Hematology parameters included basophils, eosinophils, lymphocytes, monocytes, platelet count, segmented neutrophils, total neutrophils and WBC count. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline and Week 12 in basophils, eosinophils, lymphocytes, monocytes, platelet count, segmented neutrophils, total neutrophils and WBC count are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gigacells per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Gigacells per Liter
  Basophils: number analyzed (Participants) | 80 | 71 | 72 | 76
  Basophils | -0.000 (0.0186) | 0.000 (0.0186) | 0.002 (0.0185) | -0.002 (0.0192)
  Eosinophils: number analyzed (Participants) | 80 | 71 | 72 | 76
  Eosinophils | -0.000 (0.0686) | -0.008 (0.0789) | 0.004 (0.1070) | -0.005 (0.0788)
  Lymphocytes: number analyzed (Participants) | 80 | 71 | 72 | 76
  Lymphocytes | 0.025 (0.4305) | 0.121 (0.3786) | 0.020 (0.3901) | 0.013 (0.3742)
  Monocytes: number analyzed (Participants) | 80 | 71 | 72 | 76
  Monocytes | 0.021 (0.0903) | -0.008 (0.1224) | 0.007 (0.1033) | -0.007 (0.1340)
  Platelet count: number analyzed (Participants) | 80 | 71 | 71 | 76
  Platelet count | -4.463 (28.6153) | -8.507 (28.6061) | -7.127 (33.4873) | -1.316 (53.4174)
  Segmented neutrophils: number analyzed (Participants) | 80 | 71 | 72 | 76
  Segmented neutrophils | -0.126 (0.8908) | 0.160 (0.9377) | -0.076 (1.0209) | 0.044 (0.8687)
  Total neutrophils: number analyzed (Participants) | 80 | 71 | 72 | 76
  Total neutrophils | -0.127 (0.8909) | 0.160 (0.9377) | -0.076 (1.0209) | 0.043 (0.8686)
  WBC count: number analyzed (Participants) | 80 | 71 | 72 | 76
  WBC count | -0.078 (1.1316) | 0.265 (1.0780) | -0.043 (1.1956) | 0.042 (0.9380)

23. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Albumin and Total Protein at Week 12
Description: Clinical chemistry parameters included albumin and total protein. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
Gram per Liter
  Albumin: number analyzed (Participants) | 81 | 72 | 74 | 79
  Albumin | -0.333 (2.3979) | -1.194 (1.9183) | -1.743 (2.1775) | -0.810 (2.3484)
  Total Protein: number analyzed (Participants) | 81 | 72 | 74 | 79
  Total Protein | -0.519 (3.6301) | -0.306 (3.1248) | -0.892 (3.5791) | -0.506 (3.6755)

24. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Creatinine, Direct Bilirubin, Total Bilirubin and Uric Acid at Week 12
Description: Clinical chemistry parameters included creatinine, direct bilirubin, total bilirubin and uric acid. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Micromoles per Liter
  Creatinine | -1.765 (5.5052) | 0.847 (8.3795) | 0.811 (6.6676) | -0.506 (7.1052)
  Direct bilirubin | -0.037 (0.7817) | -0.097 (0.7152) | -0.122 (0.8432) | -0.076 (0.8129)
  Total bilirubin | -0.556 (3.0083) | -0.667 (3.9611) | -1.324 (2.8579) | -0.646 (3.0215)
  Uric acid | 1.395 (41.3998) | 0.278 (42.8302) | 11.324 (40.0196) | 1.532 (37.4983)

25. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST) at Week 12
Description: Clinical chemistry parameters included ALT, ALP and AST. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Units per Liter
  ALT | 0.160 (6.8838) | -2.681 (10.3200) | -1.986 (8.8943) | -2.291 (6.9746)
  ALP | -0.037 (10.0629) | -6.403 (9.8577) | -8.878 (13.2520) | -1.962 (11.0598)
  AST | -0.247 (5.2190) | -1.139 (7.3356) | -0.743 (6.7643) | -1.228 (4.8831)

26. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Calcium, Carbon Dioxide (C02) Content, Chloride, Phosphorous, Inorganic, Potassium, Sodium and Urea at Week 12
Description: Clinical chemistry parameters included calcium, C02 content, chloride, phosphorous, inorganic, potassium, sodium and urea. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimol per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Millimol per Liter
  Calcium | -0.009 (0.0730) | -0.039 (0.0987) | -0.050 (0.0815) | -0.051 (0.0813)
  C02 content/bicarbonate | 0.728 (2.9284) | 0.014 (2.2611) | -0.486 (2.6651) | -0.506 (2.9651)
  Chloride | 0.012 (2.0946) | 0.389 (2.3887) | 0.189 (2.1433) | 0.304 (2.1204)
  Phosphorous-inorganic | 0.007 (0.2167) | -0.046 (0.1525) | -0.029 (0.3494) | -0.060 (0.1538)
  Potassium | -0.049 (0.2916) | -0.038 (0.4061) | 0.004 (0.3134) | -0.035 (0.3955)
  Sodium | -0.420 (1.8899) | 0.139 (2.0849) | -0.608 (1.7736) | -0.076 (1.7743)
  Urea | 0.102 (1.2350) | 0.160 (1.3445) | 0.385 (1.1448) | -0.097 (1.3095)

27. Secondary Outcome: Mean Change in Frequency of VMS From Baseline to Weeks 4 and 8
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an eDiary using as Global Change Question. The frequency was assessed using the question 1 as "Since you started the study medication, how has the number of your hot flashes (including night sweats) changed?". the response was rated on a 7-point scale from +3 to -3, where +3=A great deal better, +2=Moderately better, +1=A little better, 0=No change, -1=A little worse, -2=Moderately worse and -3=A great deal worse. The score ranged from +3 to -3, where +3 implied absence of symptoms and lower score implied more severe symptoms. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population with LOCF analysis. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Week 4: number analyzed (Participants) | 87 | 75 | 80 | 84
  Week 4 | -4.20 (0.435) | -3.95 (0.487) | -4.27 (0.469) | -5.68 (0.447)
  Week 8: number analyzed (Participants) | 88 | 75 | 81 | 84
  Week 8 | -5.00 (0.446) | -4.09 (0.500) | -4.07 (0.479) | -7.24 (0.459)

28. Secondary Outcome: Mean Change in Severity of VMS From Baseline to Weeks 4 and 8
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an eDiary using global change questions. The VMS severity was as follows: mild=score of 1 (brief wave of heat with minimal discomfort, usually without perspiration; able to continue activity [or sleep]), moderate=score of 2(heat with some discomfort, usually with perspiration; minimal interruption of activity [or sleep]), severe=score of 3(intense heat with considerable discomfort, usually with heavy sweating; may be unable to resume activity [or sleep] right away) and extremely severe=score of 4 (unbearable heat with intense discomfort, usually with pouring sweat; may be unable to resume activity [or sleep] for quite a while). Total score ranged from 1 to 4 and is the sum of severity scores divided by total number of VMS events. Higher score indicates worst condition. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population with LOCF analysis. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Week 4: number analyzed (Participants) | 87 | 75 | 80 | 84
  Week 4 | -0.39 (0.072) | -0.22 (0.079) | -0.22 (0.076) | -0.62 (0.073)
  Week 8: number analyzed (Participants) | 88 | 75 | 81 | 84
  Week 8 | -0.32 (0.081) | -0.11 (0.091) | -0.14 (0.086) | -0.77 (0.083)

29. Secondary Outcome: Number of Participants With VMS Percent Change From Baseline Responders With a Reduction in Frequency at Week 12 of at Least 50%, at Least 75%, and 100%
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an eDiary using global change question. The severity of VMS events were calculated using self-reported participants assessments recorded and transmitted by eDiary. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Percent change was calculated by multiplying the change from baseline value with 100. Number of participants with VMS percent change from Baseline responders with a reduction in frequency at Week 12 of at least 50%, at least 75%, and 100% are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF analysis. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 88 | 75 | 81 | 84
Participants
  At least 50% reduction in frequency | 43 | 36 | 32 | 61
  At least 75% reduction in frequency | 21 | 16 | 15 | 42
  At least 100% reduction in frequency | 3 | 1 | 0 | 10

30. Secondary Outcome: Number of Participants With VMS Percent Change From Baseline Responders With a Reduction in Severity at Week 12 of at Least 50%, at Least 75%, and 100%
Description: Individual VMS (hot flash or night sweats) events were recorded by participants in an eDiary using global change questions. The VMS severity was as follows: mild (brief wave of heat with minimal discomfort, usually without perspiration; able to continue activity [or sleep]), moderate (heat with some discomfort, usually with perspiration; minimal interruption of activity [or sleep]), severe (intense heat with considerable discomfort, usually with heavy sweating; may be unable to resume activity [or sleep] right away) and extremely severe (unbearable heat with intense discomfort, usually with pouring sweat; may be unable to resume activity [or sleep] for quite a while). The severity of VMS events were calculated using self-reported participants assessments recorded and transmitted by eDiary. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Percent change was calculated by multiplying change from Baseline value with 100.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF analysis. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 88 | 75 | 81 | 84
Participants
  At least 50% reduction in severity | 8 | 7 | 3 | 28
  At least 75% reduction in severity | 3 | 1 | 0 | 10
  At least 100% reduction in severity | 3 | 1 | 0 | 10

31. Secondary Outcome: Change in Menopause Quality of Life (MENQoL) Score From Baseline to Visits 6 (Week 4) and Visit 8 (Week 12)
Description: MENQOL instrument is a 32-item, validated questionnaire designed to measure symptoms that participants experience due to menopause and degree to which these symptoms bother them. Each item references a symptom and is composed of two-part question; a yes/no confirmation that the participant has symptom followed by a question asking how bothersome the symptom is, if present. The MENQOL items are designed to be grouped into domains that address vasomotor (items 1-3), psychosocial(items 4-10), physical (items 11-26, 30-32) and sexual symptoms (items 27-29). Each domain is given a separate score; there is no overall score. The domain score is sum of individual item scores divided by number of items in that domain. Since domain subscales are not comprised of an equivalent number of items, mean of subscale is used as overall subscale score. Each domain score ranges from 1 to 8. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Vasomotor Domain Score; Week 4: number analyzed (Participants) | 83 | 71 | 79 | 79
  Vasomotor Domain Score; Week 4 | -1.36 (0.205) | -1.26 (0.227) | -1.27 (0.213) | -2.13 (0.207)
  Psychosocial Domain Score; Week 4: number analyzed (Participants) | 82 | 70 | 78 | 76
  Psychosocial Domain Score; Week 4 | -0.51 (0.157) | -0.46 (0.173) | -0.42 (0.165) | -0.63 (0.161)
  Physical Domain Score; Week 4: number analyzed (Participants) | 82 | 70 | 77 | 78
  Physical Domain Score; Week 4 | -0.65 (0.122) | -0.50 (0.135) | -0.58 (0.127) | -0.70 (0.123)
  Sexual Domain Score; Week 4: number analyzed (Participants) | 79 | 71 | 73 | 76
  Sexual Domain Score; Week 4 | -0.62 (0.187) | -0.62 (0.203) | -0.62 (0.200) | -0.85 (0.188)
  Vasomotor Domain Score; Week 12: number analyzed (Participants) | 81 | 75 | 76 | 84
  Vasomotor Domain Score; Week 12 | -1.79 (0.241) | -1.21 (0.260) | -1.09 (0.253) | -2.99 (0.237)
  Psychosocial Domain Score; Week 12: number analyzed (Participants) | 80 | 72 | 75 | 85
  Psychosocial Domain Score; Week 12 | -0.46 (0.178) | -0.45 (0.193) | -0.33 (0.189) | -0.91 (0.174)
  Physical Domain Score; Week 12: number analyzed (Participants) | 80 | 73 | 75 | 85
  Physical Domain Score; Week 12 | -0.59 (0.133) | -0.36 (0.144) | -0.50 (0.139) | -0.87 (0.129)
  Sexual Domain Score; Week 12: number analyzed (Participants) | 81 | 72 | 72 | 83
  Sexual Domain Score; Week 12 | -0.47 (0.194) | -0.18 (0.214) | -0.52 (0.215) | -1.04 (0.194)

32. Secondary Outcome: Change in Medical Outcomes Study (MOS) Sleep Score From Baseline to Visits 6 (Week 4) and Visit 8 (Week 12)
Description: The MOS Sleep Scale is a validated questionnaire designed to measure a participant sleep quality via 12 questions. Items are designed to be grouped into domains that include sleep disturbance (items 1, 3, 7, 8), sleep adequacy (items 4, 12), daytime somnolence (items 6, 9, 11), sleep quantity (2), 6-Item Sleep Scale (items 4, 5, 7, 8, 9, 12) and 9-Item Sleep Scale (items 3, 4, 5, 6, 7, 8, 9, 11, 12). Each domain is given a separate score. The domain score is calculated as the sum of the individual item scores in that domain. Transformed scores were calculated for the domains only. This transformation converts the raw domain score to a 0 to 100 scale following the formula: Transformed score = ([Raw score - Lowest possible score]/Possible score range)*100. Lowest score 0 indicates best sleep quality and higher score 100 indicates worst sleep quality. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Sleep Disturbance domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 84
  Sleep Disturbance domain; Week 4 | 1.62 (0.378) | 1.29 (0.422) | 1.05 (0.400) | 1.68 (0.386)
  Sleep Adequacy domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Sleep Adequacy domain; Week 4 | 0.57 (0.294) | 0.66 (0.329) | 0.37 (0.311) | 1.00 (0.300)
  Sleep Somnolence domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Sleep Somnolence domain; Week 4 | 0.43 (0.297) | -0.19 (0.332) | 0.00 (0.314) | 0.65 (0.303)
  Sleep Quantity domain; Week 4: number analyzed (Participants) | 72 | 64 | 70 | 72
  Sleep Quantity domain; Week 4 | 0.24 (0.121) | 0.21 (0.134) | 0.13 (0.127) | 0.47 (0.124)
  6-Item Sleep Scale domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  6-Item Sleep Scale domain; Week 4 | 2.19 (0.560) | 1.85 (0.621) | 1.53 (0.588) | 2.87 (0.568)
  9-Item Sleep Scale domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  9-Item Sleep Scale domain; Week 4 | 3.01 (0.774) | 2.26 (0.858) | 2.01 (0.813) | 4.05 (0.784)
  Transformed Sleep Disturbance domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Transformed Sleep Disturbance domain; Week 4 | 6.76 (1.577) | 5.35 (1.758) | 4.37 (1.667) | 7.01 (1.607)
  Transformed Sleep Adequacy domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Transformed Sleep Adequacy domain; Week 4 | 4.75 (2.450) | 5.48 (2.738) | 3.10 (2.594) | 8.35 (2.501)
  Transformed Sleep Somnolence domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Transformed Sleep Somnolence domain; Week 4 | 2.38 (1.651) | -1.03 (1.842) | 0.02 (1.747) | 3.62 (1.685)
  Transformed 6-Item Sleep Scale domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Transformed 6-Item Sleep Scale domain; Week 4 | 6.08 (1.556) | 5.15 (1.724) | 4.25 (1.634) | 7.98 (1.577)
  Transformed 9-Item Sleep Scale domain; Week 4: number analyzed (Participants) | 84 | 73 | 79 | 80
  Transformed 9-Item Sleep Scale domain; Week 4 | 5.57 (1.434) | 4.19 (1.588) | 3.73 (1.506) | 7.50 (1.453)
  Sleep Disturbance domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Sleep Disturbance domain; Week 12 | 1.34 (0.366) | 1.37 (0.397) | 0.82 (0.390) | 2.12 (0.364)
  Sleep Adequacy domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Sleep Adequacy domain; Week 12 | 1.36 (0.302) | 0.79 (0.328) | 0.02 (0.322) | 1.36 (0.301)
  Sleep Somnolence domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Sleep Somnolence domain; Week 12 | 0.07 (0.295) | 0.41 (0.321) | 0.13 (0.315) | 1.17 (0.294)
  Sleep Quantity domain; Week 12: number analyzed (Participants) | 72 | 69 | 63 | 75
  Sleep Quantity domain; Week 12 | 0.22 (0.131) | 0.23 (0.142) | -0.08 (0.142) | 0.46 (0.133)
  6-Item Sleep Scale domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  6-Item Sleep Scale domain; Week 12 | 2.62 (0.571) | 2.19 (0.616) | 0.57 (0.604) | 3.68 (0.565)
  9-Item Sleep Scale domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  9-Item Sleep Scale domain; Week 12 | 2.87 (0.774) | 3.17 (0.834) | 1.36 (0.818) | 5.32 (0.765)
  Transformed Sleep Disturbance domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Transformed Sleep Disturbance domain; Week 12 | 5.57 (1.525) | 5.70 (1.654) | 3.41 (1.627) | 8.85 (1.518)
  Transformed Sleep Adequacy domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Transformed Sleep Adequacy domain; Week 12 | 11.35 (2.514) | 6.62 (2.734) | 0.19 (2.682) | 11.30 (2.508)
  Transformed Sleep Somnolence domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Transformed Sleep Somnolence domain; Week 12 | 0.41 (1.639) | 2.30 (1.781) | 0.72 (1.749) | 6.48 (1.635)
  Transformed 6-Item Sleep Scale domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Transformed 6-Item Sleep Scale domain; Week 12 | 7.27 (1.586) | 6.08 (1.711) | 1.57 (1.678) | 10.23 (1.570)
  Transformed 9-Item Sleep Scale domain; Week 12: number analyzed (Participants) | 83 | 78 | 76 | 85
  Transformed 9-Item Sleep Scale domain; Week 12 | 5.32 (1.433) | 5.88 (1.544) | 2.51 (1.515) | 9.85 (1.417)

33. Secondary Outcome: Changes in Vulvar Vaginal Atrophy (VVA) Symptom Score From Baseline to Visit 8 (Week 12)
Description: The VVA Symptoms Scale questionnaire is an 18-item instrument that captures symptoms related to VVA, asks participant to identify symptom that bothers them the most and contains items to assess degree of bother participants experience from each symptom and impact that most bothersome symptom has on their daily life. Items 1 to 8 had responses and scores of none=0, mild=1, moderate=2 and severe=3. Items 9 to 18 had responses and scores of not at all=0, a little=1, moderately=2 and a lot=3. Severity item and bothersome item respectively were as follows: vaginal dryness:1 and 9; Vaginal itching:2 and 10; Vaginal irritation:3 and 11; Painful urination:4 and 12; Difficulty urinating:5 and 13; Vaginal pain associated with sexual activity:6 and 14; Vaginal bleeding associated with sexual activity:7 and 15. Total score ranged from 0 to 3; higher score indicated most bothersome. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) to Visit 8 (Week 12)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Severity of vaginal dryness: number analyzed (Participants) | 83 | 78 | 76 | 85
  Severity of vaginal dryness | -0.2 (0.79) | -0.1 (0.81) | -0.3 (0.86) | -0.4 (1.03)
  Severity of vaginal itching: number analyzed (Participants) | 83 | 78 | 75 | 85
  Severity of vaginal itching | 0.0 (0.75) | 0.1 (0.65) | -0.2 (0.74) | 0.0 (0.58)
  Severity of vaginal irritation: number analyzed (Participants) | 83 | 78 | 76 | 85
  Severity of vaginal irritation | 0.0 (0.65) | 0.0 (0.50) | -0.1 (0.74) | 0.0 (0.67)
  Severity of painful urination: number analyzed (Participants) | 83 | 78 | 76 | 85
  Severity of painful urination | 0.0 (0.43) | 0.0 (0.36) | 0.0 (0.48) | -0.1 (0.64)
  Severity of urinating difficulty: number analyzed (Participants) | 83 | 78 | 76 | 85
  Severity of urinating difficulty | 0.0 (0.19) | 0.0 (0.43) | -0.1 (0.36) | 0.0 (0.50)
  Severity of vaginal pain due to sexual activity: number analyzed (Participants) | 81 | 75 | 71 | 84
  Severity of vaginal pain due to sexual activity | -0.1 (0.75) | 0.0 (0.78) | -0.1 (0.93) | -0.4 (0.98)
  Vaginal bleeding severity due to sexual activity: number analyzed (Participants) | 82 | 75 | 71 | 84
  Vaginal bleeding severity due to sexual activity | 0.0 (0.00) | 0.0 (0.35) | 0.0 (0.36) | 0.0 (0.15)
  Bothered by vaginal dryness: number analyzed (Participants) | 57 | 58 | 62 | 63
  Bothered by vaginal dryness | -0.1 (0.79) | -0.1 (0.83) | -0.3 (0.89) | -0.3 (1.04)
  Bothered by vaginal itching: number analyzed (Participants) | 58 | 57 | 62 | 59
  Bothered by vaginal itching | -0.1 (0.69) | 0.0 (0.58) | -0.3 (0.72) | 0.1 (0.69)
  Bothered by vaginal irritation: number analyzed (Participants) | 57 | 57 | 62 | 59
  Bothered by vaginal irritation | -0.1 (0.74) | -0.1 (0.66) | -0.2 (0.77) | -0.1 (0.63)
  Bothered by painful urination: number analyzed (Participants) | 57 | 57 | 63 | 62
  Bothered by painful urination | -0.1 (0.48) | 0.1 (0.46) | -0.1 (0.69) | -0.1 (0.52)
  Bothered by difficulty in urination: number analyzed (Participants) | 57 | 57 | 62 | 63
  Bothered by difficulty in urination | -0.1 (0.34) | 0.1 (0.40) | -0.1 (0.51) | 0.0 (0.46)
  Bothered by vaginal pain due to sexual activity: number analyzed (Participants) | 57 | 56 | 59 | 61
  Bothered by vaginal pain due to sexual activity | -0.2 (0.84) | -0.1 (0.70) | 0.0 (0.96) | -0.3 (0.95)
  Vaginal bleeding due to sexual activity bothering: number analyzed (Participants) | 57 | 54 | 59 | 59
  Vaginal bleeding due to sexual activity bothering | 0.0 (0.00) | 0.0 (0.41) | -0.1 (0.58) | 0.0 (0.13)
  Vaginal symptoms interference with sexual activity: number analyzed (Participants) | 58 | 55 | 60 | 66
  Vaginal symptoms interference with sexual activity | -0.1 (0.85) | -0.1 (0.86) | -0.2 (1.10) | -0.6 (1.15)
  Vaginal symptoms interference with social activity: number analyzed (Participants) | 59 | 57 | 62 | 66
  Vaginal symptoms interference with social activity | 0.0 (0.69) | -0.1 (0.62) | -0.1 (0.88) | -0.2 (0.72)
  Vaginal symptoms interference with daily activity: number analyzed (Participants) | 58 | 57 | 63 | 67
  Vaginal symptoms interference with daily activity | -0.1 (0.80) | 0.0 (0.50) | -0.2 (0.64) | -0.2 (0.57)

34. Secondary Outcome: Change in Brief Fatigue Inventory (BFI) Score From Visit 2 to Visit 7
Description: The BFI is a validated questionnaire designed to measure a participant's fatigue via nine questions that are summated to create a total score. Items 1-3 request a rating on a scale ranging from 0 - 10 with 0 representing 'No Fatigue' and 10 representing 'As bad as you can imagine'. Five items 4A-4F request an interference score on a scale ranging from 0 - 10 with 0 representing 'Does not interfere' and 10 representing 'Completely Interferes'. The values of the scales for all items was used in scoring the response to each item. The following groupings of items was used to create domain scores. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. Higher score indicates more severe fatigue. Visit 2 was Day -21. Change from Visit 2 was calculated by subtracting Visit 2 values from post-Visit 2 values.
Time Frame: Visit 2 (Day -21) to Visit 7 (Week 8)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Total Score: number analyzed (Participants) | 82 | 71 | 74 | 77
  Total Score | -0.84 (0.251) | -0.43 (0.279) | -0.33 (0.270) | -0.40 (0.260)
  Severity domain: number analyzed (Participants) | 82 | 70 | 74 | 76
  Severity domain | -0.87 (0.289) | -0.58 (0.323) | -0.53 (0.314) | -0.43 (0.301)
  Interference domain: number analyzed (Participants) | 82 | 71 | 74 | 77
  Interference domain | -0.82 (0.261) | -0.33 (0.290) | -0.25 (0.281) | -0.38 (0.271)

35. Secondary Outcome: Change in the Centers for Epidemiologic Studies in Depression (CES-D) Score From Visit 2 to Visit 7
Description: The CES-D is a questionnaire designed to measure depressive symptoms via 20 items that are summed to create a total score. Depressive symptoms are fairly common in postmenopausal women, and it's possible that stimulation of estrogen receptors via a selective estrogen receptor modulator may improve depressive symptoms. Questions 4, 8, 12 and 16 are weighted negatively (the scores are flipped prior to creating total score). If 3 or more items are missing then total score is missing. If fewer than 3 items are missing then missing item is set to group mean of that item for appropriate randomized treatment group. These means are only calculated if more than half of the participants used for calculation have responded to item. The items are summed to give total score ranging from 0 to 60. Lower score 0=no depression, higher score 60=higher degree of depression severity. Visit 2 was Day -21. Change from Visit 2 was calculated by subtracting Visit 2 values from post-Visit 2 values.
Time Frame: Visit 2 (Day -21) to Visit 7 (Week 8)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 78 | 70 | 74 | 77
Scores on a Scale | -2.55 (1.077) | -1.26 (1.172) | -0.38 (1.132) | -1.27 (1.090)

36. Secondary Outcome: Change in Work Productivity and Activity Impairment (WPAI) Score From Visit 2 to Visit 7
Description: The WPAI is a questionnaire that measured workplace productivity and absenteeism via 6 items/questions, adapted to participants experiencing menopausal symptoms. Item 1 asks about current employment with a yes/no response. Items 2- 4 ask for continuous response in hours. Item 5 asks for response on rating scale related to WP ranging from 0:Menopausal symptoms had no effect on work to 10:Couldn't work at all. Item 6 asks for response on rating scale related to daily activities ranging from 0:no effect on daily activities to 10:Couldn't perform any daily activities. The score calculation- Effect on work: (Item 5 score÷10); Absenteeism: (Item 2÷Item 2+Item 4); Overall work impairment ([Item 2÷Item 2+Item 4]+ [1- {Item 2÷Item 2+Item 4}]*[ Item 5 score÷10]); Activity impairment: (Item 6 score÷10). Total score range from 0 to 10 where higher score indicates worst condition. Visit 2 was Day -21. Change from Visit 2 was calculated by subtracting Visit 2 values from post-Visit 2 values.
Time Frame: Visit 2 (Day -21) to Visit 7 (Week 8)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 89 | 90
Scores on a Scale
  Effect on work: number analyzed (Participants) | 55 | 45 | 50 | 44
  Effect on work | -16.80 (3.319) | -11.71 (3.681) | -6.43 (3.199) | -17.69 (3.437)
  Absenteeism: number analyzed (Participants) | 48 | 35 | 38 | 38
  Absenteeism | -1.10 (1.229) | -2.01 (1.409) | -2.67 (1.224) | -0.51 (1.211)
  Overall work impairment: number analyzed (Participants) | 48 | 35 | 38 | 37
  Overall work impairment | -19.37 (3.761) | -17.82 (4.318) | -13.30 (3.768) | -18.48 (3.763)
  Activity impairment: number analyzed (Participants) | 79 | 71 | 74 | 77
  Activity impairment | -20.21 (2.823) | -13.50 (3.082) | -7.57 (2.972) | -18.58 (2.886)

37. Secondary Outcome: Change From Visit 2 to Visit 8 in Vaginal pH
Description: Vaginal pH was measured at Visit 2 and Visit 8 using standard pH indicator strips available at the participating site clinic. The pH indicator strip was inserted to the upper portion of the proximal one third of the vaginal vault, placed in contact with the lateral vaginal mucosal wall for approximately 1 minute, and evaluated according to the instructions provided in the package labeling. pH is calculated on a scale of 0 to 14, such that, the lower the number, more acidic the vagina and higher the number, more alkaline the vagina with 7 being neutral. Change from Visit 2 to Visit 8 was calculated by subtracting Visit 2 values from Visit 8 values.
Time Frame: Visit 2 (Day -21) to Visit 8 (Week 12)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 74 | 75 | 84
Points on a scale | -0.13 (0.137) | -0.03 (0.151) | -0.09 (0.146) | -0.59 (0.138)

38. Secondary Outcome: Change From Visit 2 to Visit 8 in Percentage of Superficial Cells to Determine the Vaginal Maturation Index (VMI)
Description: A lateral vaginal wall specimen was collected at Visit 2 (Day -21) and Visit 8 (Week 12) and was sent to Central Pathology for analysis. Parabasal, intermediate, and superficial squamous cells were counted and percentages calculated. The VMI (also referred to as Maturation Value [MV]) of the vaginal mucosa was calculated according to the following equation:
  VMI (MV)= (% Intermediate Cells x 0.5) + (% Superficial cells). Visit 2 was Day -21 and Visit 8 was Week 12. Change from Visit 2 to Visit 8 was calculated by subtracting Visit 2 values from Visit 8 values.
Time Frame: Visit 2 (Day -21) to Visit 8 (Week 12)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of cells
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 68 | 61 | 64 | 69
Percentage of cells | -1.0 (1.99) | -0.3 (2.16) | 9.2 (2.11) | 13.5 (2.05)

39. Secondary Outcome: Change From Baseline in Glucose at Week 12
Description: Pharmacodynamic marker included glucose. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Millimoles per Liter | 0.119 (0.7004) | 0.078 (0.6010) | -0.072 (0.7097) | -0.110 (0.6488)

40. Secondary Outcome: Change From Baseline at Week 12 in Serum Hormone Levels- Estradiol
Description: Serum hormone included Estradiol. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline at Week 12 in estradiol are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 80 | 71 | 72 | 77
Picomoles per Liter | -1.775 (88.9767) | 2.324 (71.5970) | -8.403 (120.9173) | 178.312 (618.0547)

41. Secondary Outcome: Change From Baseline at Week 12 in Serum Hormone Levels- Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: Serum hormones included FSH and LH. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 90 | 87 | 88 | 90
International units per Liter
  FSH: number analyzed (Participants) | 81 | 72 | 74 | 79
  FSH | 0.359 (12.4050) | -5.322 (15.3625) | -7.999 (17.5791) | -18.401 (18.6976)
  LH: number analyzed (Participants) | 81 | 72 | 74 | 79
  LH | -1.454 (9.7558) | -1.571 (8.6063) | -3.362 (9.4806) | -1.732 (13.2826)

42. Secondary Outcome: Change From Baseline at Week 12 in Serum Hormone Levels- Testosterone
Description: Serum hormones included testosterone. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. Mean change from Baseline at Week 12 in testosterone are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomol per Liter
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Nanomol per Liter | -0.086 (0.5454) | 0.115 (0.5598) | 0.105 (0.4587) | -0.009 (0.4252)

43. Secondary Outcome: Change From Baseline at Week 12 in Waist Circumference
Description: To measure waist circumference, clothing was lifted from around the waist to ensure correct positioning of the measuring tape. Participants were instructed to stand erect with abdomen relaxed, arms at side, feet together, and weight equally divided over both legs. The non-stretchable tape was placed at the waist midway between the palpated iliac crest and the palpated lowest rib margin in the left and right mid-axillary lines. The tape was even, parallel to the floor not twisted with the measurement scale facing outward. The assessor was instructed to ensure that the tape was just touching the skin but not compressing the soft tissue. The measurement was made at the end of a normal expiration. The waist was measured at least twice or more if necessary, until two measurements were within 1 centimeter and the confirmatory reading recorded to one decimal place. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Centimeters | -0.83 (0.651) | -1.29 (0.728) | 1.03 (0.709) | 0.12 (0.680)

44. Secondary Outcome: Change From Baseline at Week 12 in Hip Circumference
Description: For hip circumference, the participant was instructed to stand erect with arms at sides and feet together. The measurement was taken at the point yielding the maximum circumference over the buttocks (widest part of the greater trochanters) with nonstretchable tape. The tape was even, not twisted with the measurement scale facing outward. The assessor was instructed to ensure that the tape was just touching the skin but not compressing the soft tissue. The hip should be measured at least twice until two measurements are within 1 centimeter and the last reading recorded. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 73 | 79
Centimeters | -0.72 (0.596) | 0.13 (0.666) | 0.89 (0.650) | 0.14 (0.621)

45. Secondary Outcome: Change From Baseline at Week 12 in Weight
Description: Participants were weighed on a calibrated balance beam or digital scale. Participants were instructed to be dressed in light indoor clothing without shoes and also to have empty pockets and to void before weighing. It was strongly recommended that participants were weighed in the morning at the beginning of the clinic visit. Weight was measured at least twice or more if necessary, until two measurements were within 0.5 kilograms. The last (confirmed) reading was recorded in the electronic case report form. Weight was recorded in kilograms to the nearest tenth. When the weight was measured in pounds, it was converted into kilograms using the conversion factor: pounds/ 2.2 = kilograms. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Kilograms | 0.13 (0.224) | 0.38 (0.250) | 0.36 (0.243) | 0.64 (0.234)

46. Secondary Outcome: Change From Baseline at Week 12 in Body Mass Index (BMI)
Description: BMI was calculated from height (taken at Screening Visit 1 [Day -35]) and weight at Week 12 using the formula: BMI = [weight in kilograms divided by (height in meters)^2]. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Kilogram per square meters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 81 | 72 | 74 | 79
Kilogram per square meters | 0.05 (0.085) | 0.15 (0.095) | 0.12 (0.092) | 0.25 (0.088)

47. Secondary Outcome: Change From Baseline at Week 12 in Abdomen Body Circumference, Abdomen Saggital Diameter and Thigh Circumference
Description: Thigh circumference was measured on the left leg directly below the gluteal fold; with the participant standing with both arms at the side, feet together, and with equal weight on both feet when this measurement was taken. The thigh was measured at least twice until two measurements were within 1 centimeter, and the last reading recorded. Abdomen body circumference and abdomen saggital diameter was measured in centimeter to once decimal place by Computerized tomography (CT) scan with the participant in supine position. CT scan of the abdomen was conducted at the Lumbar 4 vertebrae level. Scans were performed with 120 kilovolts, 5 millimeter slice thickness and 48 centimeter scan field of view. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Body Composition Population which comprised of any ITT participants who provided consent for the body composition sub-study and received additional body composition assessments. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3
Centimeters
  Abdomen body circumference | -1.20 (2.963) | -0.30 (1.739) | 2.07 (3.066) | -1.90 (2.884)
  Abdomen saggital circumference | -0.50 (1.236) | -0.04 (0.841) | 0.17 (0.379) | -0.77 (1.002)
  Thigh circumference | 0.13 (0.150) | 0.00 (0.797) | 0.23 (0.961) | -0.07 (2.250)

48. Secondary Outcome: Change From Baseline at Week 12 in Abdomen Visceral Adipose Tissue (AVAT), Abdomen Subcutaneous Adipose Tissue (ASAT), Thigh Subcutaneous Adipose Tissue (TSAT) and Thigh Intermuscular Adipose Tissue (TIAT)
Description: AVAT, ASAT, TSAT and TIAT was measured in centimeter to once decimal place by CT scan. A CT scan of the abdomen was conducted at the Lumbar 4 vertebrae level. A CT scan of the right thigh was performed at half the distance between the knee joint and greater trochanter femoralis. Scans were performed with 120 kilovolts, 5 millimeter slice thickness (thigh scan 3 millimeter slice thickness) and 48 centimeter scan field of view. Baseline was Week 0. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Week 0) and Week 12
Population: Body Composition Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Square centimeters
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
Number analyzed (Participants) | 5 | 5 | 4 | 3
Square centimeters
  AVAT: number analyzed (Participants) | 4 | 5 | 3 | 3
  AVAT | 0.50 (23.779) | 7.66 (11.251) | -5.50 (12.418) | 2.98 (5.047)
  ASAT: number analyzed (Participants) | 4 | 5 | 3 | 3
  ASAT | -3.12 (6.544) | -2.10 (18.822) | 22.37 (43.273) | -13.42 (17.175)
  TSAT: number analyzed (Participants) | 4 | 5 | 3 | 3
  TSAT | 0.73 (4.366) | 1.59 (7.763) | 6.12 (7.869) | 2.90 (13.194)
  TIAT: number analyzed (Participants) | 4 | 5 | 3 | 3
  TIAT | 0.05 (0.131) | 0.12 (0.399) | 0.18 (0.320) | 0.17 (0.322)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks.
Description: Safety Population was used.
Arm/Group | Placebo | GSK232802 25 mg | GSK232802 75 mg | Premarin 0.3 mg
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/87 | 0/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 2/90 | 0/878 | 1/88 | 1/90
Other Adverse Events (participants affected / at risk) | 30/90 | 24/87 | 21/88 | 17/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | GSK232802 25 mg (N=878) | GSK232802 75 mg (N=88) | Premarin 0.3 mg (N=90)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | GSK232802 25 mg (N=87) | GSK232802 75 mg (N=88) | Premarin 0.3 mg (N=90)
Nasopharyngitis (Infections and infestations) | 8 | 3 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 3 | 3
Nausea (Gastrointestinal disorders) | 5 | 6 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 4 | 3
Headache (Nervous system disorders) | 14 | 8 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.